CLINICAL TRIAL: NCT01184833
Title: Evaluation of Risk Factors for Premature Discontinuation of Injection Treatment With Betaferon in Patients With Relapsing Forms of Multiple Sclerosis
Brief Title: Evaluation of Risk Factors for Early Termination of Injection Treatment With Betaferon in Patients Suffering From Multiple Sclerosis
Acronym: BREAK
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Medical Director, Bayer Sp. z o.o.
Other Study IDs: 14323; BF0813PL (Other: company internal)
Record Dates: First submitted 2010-08-18; First posted 2010-08-19 (Estimated); Last update posted 2013-06-25 (Estimated); Status verified 2013-06

CONDITIONS: Multiple Sclerosis
Keywords: Multiple sclerosis; Interferon beta-1b; Compliance to treatment; Premature treatment discontinuation
MeSH Terms: conditions — Multiple Sclerosis | interventions — Interferon beta-1b

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1
  Interventions: Drug: Interferon beta-1b (Betaseron, BAY86-5046)

INTERVENTIONS:
Drug: Interferon beta-1b (Betaseron, BAY86-5046) — Patients treated with regular dose of Betaferon injections (250 micrograms subcutaneously every other day) under the routine practice setting.

SUMMARY:
Non-adherence to the treatment regimen is a common problem associated with injectable drugs (e.g. Betaferon) that are used in multiple sclerosis patients.

Certain patients omit single injections or even totally discontinue therapy that normally should be long-term. It is therefore crucial to identify the factors which have the most significant effect on regularity of administration of Betaferon and the risk of premature discontinuation of treatment in order to undertake appropriate preventive measures.

This study is conducted in routine practice setting and aims to identify those risks. Pre-defined risk factors associated with technical aspects of the treatment, support provided to the patient, stage of the disease and possible adverse effects of the medication are checked on a quarterly basis with a questionnaire method. Monitoring of omitted doses of the prescribed medication (Betaferon) is carried out by the study nurse.

ELIGIBILITY:
Inclusion Criteria:

* Relapsing-remitting multiple sclerosis
* Age >/= 18 years
* Start of treatment with Betaferon not earlier than 60 days prior to inclusion

Exclusion Criteria:

* Synonymous with contraindications to Betaferon

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with relapsing form of multiple sclerosis treated with Betaferon under routine practice setting.
Sampling Method: Probability Sample
Enrollment: 852 (Actual)
Dates: Start 2008-09; Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Rate of discontinuation of Betaferon | 24 months

SECONDARY OUTCOMES:
Number of missed doses of Betaferon | 24 months
Depression score as measured by CES-D questionnaire | 24 months
Neurological disability score as measured by EDSS scale | 24 months
Overall tolerability of treatment as measured by rate of adverse events | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Many Locations, Poland